CLINICAL TRIAL: NCT05813847
Title: A Randomized, Double-Blind, Placebo- and Active-Controlled Study to Evaluate the Efficacy and Safety of CPL-01 in the Management of Postoperative Pain After Open Inguinal Herniorrhaphy
Brief Title: Herniorrhaphy for Postoperative Pain
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cali Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPL-01-301
Record Dates: First submitted 2023-04-03; First posted 2023-04-14 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Hernia, Inguinal
MeSH Terms: conditions — Hernia, Inguinal | interventions — Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CPL-01 (Experimental): Local infiltration of CPL-01
  Interventions: Drug: local anaesthetic injection
- Ropivacaine HCl (Active Comparator): Local infiltration of Naropin
  Interventions: Drug: local anaesthetic injection
- Placebo (Placebo Comparator): Local infiltration of Saline Placebo
  Interventions: Drug: local anaesthetic injection

INTERVENTIONS:
Drug: local anaesthetic injection — Local infiltration of study drug

SUMMARY:
Subjects receive either CPL-01, positive control, or negative control after herniorrhaphy and are then followed.

ELIGIBILITY:
Inclusion Criteria:

* Able to sign Informed Consent
* Scheduled to have inguinal hernia repair
* Be a reasonably healthy adult 18 - 75 years of age
* Body mass index ≤ 39 kg/m2
* If biologically female, not pregnant or planning to become pregnant
* If biologically male, using acceptable birth control
* Be willing and able to complete study procedures

Exclusion Criteria:

* Previously inguinal herniorrhaphy
* Concurrent painful condition that may require analgesic treatment
* History or clinical manifestation of significant medical, neuropsychiatric, or other condition, significant abnormal clinical laboratory test value, or known bleeding abnormality that could preclude or impair study participation
* Clinically significant existing arrhythmia, bundle branch block or abnormal ECG, myocardial infarction, or coronary arterial bypass graft surgery within the prior 12 months
* History of malignant hyperthermia or glucose-6-phosphate dehydrogenase deficiency.
* Impaired liver function (e.g., alanine aminotransferase [ALT] > 3 × upper limit of normal [ULN] or total bilirubin > 2 × ULN), active hepatic disease, or cirrhosis.
* Impaired renal function (e.g., creatinine > 1.5 × ULN).
* Malignancy in the past year
* Known or suspected daily use of opioids for 7 or more consecutive days within the previous 6 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain control | 72 hours
  Area under the curve of the numeric rating score for pain with activity, where 0 is no pain and 10 is worst pain imaginable

CONTACTS AND LOCATIONS:
Overall Officials: Erol Onel, Study Director — Cali Biosciences
Locations (1):
- Todd Bertoch, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No